CLINICAL TRIAL: NCT03573934
Title: Investigation of GLP-2 Mechanism of Action (KS-2)
Brief Title: Gut Hormones and Bone Remodeling in Humans (KS-2)
Acronym: KS-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Kirsa Skov-Jeppesen, Principal Investigator., University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UCHP-KS-2
Record Dates: First submitted 2018-06-07; First posted 2018-06-29 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GLP-2 (Experimental): Glucagon-Like Peptide-2 (GLP-2) injection
  Interventions: Other: GLP-2
- GIP (Experimental): Glucose-dependent Insulinotropic polypeptide (GIP) injection
  Interventions: Other: GIP
- GLP-2+GIP (Experimental): GLP-2+GIP injection
  Interventions: Other: GLP-2+GIP
- Placebo (Placebo Comparator): Placebo injection
  Interventions: Other: Placebo

INTERVENTIONS:
Other: GLP-2 — GLP-2
  Arms: GLP-2
Other: GIP — GIP
  Arms: GIP
Other: GLP-2+GIP — GLP-2+GIP
  Arms: GLP-2+GIP
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Effects of GLP-2 and GIP on bone remodeling in healthy young men.

DETAILED DESCRIPTION:
We will investigate acute effects of GLP-2 and GIP on bone remodeling in healthy young men.

ELIGIBILITY:
Inclusion Criteria:

Age between 20 and 40 years old Caucasian Healthy BMI between 18.5 and 24.9 kg/m2.

Exclusion Criteria:

Chronic disease Smoking Medication Weight change more than 3 kg whitin the last 3 months Overweight surgery Intestinal surgery Hgb<8,0 mmol/L Decreased renal function.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Bone resorption | From -10 minutes to 240 minutes.
  C-terminal telopeptide (CTX) is a marker of bone resorption. Measured in serum.
Bone formation | From -10 minutes to 240 minutes.
  P1NP is a marker of bone formation. Measured in serum.

SECONDARY OUTCOMES:
Parathyroid hormone | From -10 minutes to 240 minutes.
  PTH is a bone marker
Calcium | From -10 minutes to 240 minutes.
  Measured in serum.
GIP | From -10 minutes to 240 minutes.
  Intact and total GIP.
GLP-2 | From -10 minutes to 240 minutes.
  Intact GLP-2
Glucose | From -10 minutes to 240 minutes.
  Measured in serum.
Insulin | From -10 minutes to 240 minutes.
  Measured in serum.
C-peptide | From -10 minutes to 240 minutes.
  Measured in serum.
Sclerostin | From -10 minutes to 240 minutes.
  Bone marker.

OTHER OUTCOMES:
Heart rate | From -10 minutes to 240 minutes.
  Before blood sampling
Blood pressure | From -10 minutes to 240 minutes.
  Before blood sampling

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided